CLINICAL TRIAL: NCT05701397
Title: Prevalence of Cardiac Amyloidosis in Patients Undergoing Surgery for Lumbar Spinal Stenosis.
Acronym: CASS-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Professor, PhD, DMSci, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1-10-72-116-22
Record Dates: First submitted 2023-01-16; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Amyloidosis; Spinal Stenosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Spinal Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients undergoing surgery for lumbar spinal stenosis. Patients will have a biopsy taken from the ligamentum flavum and test for the presence of amyloid. Patients with amyloid in the ligamentum flavum will be referred for a DPD scintigraphy.
  Interventions: Diagnostic Test: DPD scintigraphy

INTERVENTIONS:
Diagnostic Test: DPD scintigraphy — Bone tracer scintigraphy, diagnostic for transthyretin cardiac amyloidsis

SUMMARY:
Patients undergoing surgery for lumbar spinal stenosis will have biopsies of the ligamentum flavum sent to the department of pathology for histologic screening.

If the ligament biopsy contains amyloid, patients will receive an echocardiogram, an ecg, biomarker testing, and a bone tracer scintigraphy diagnostic of cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgery for lumbar spinal stenosis
* Age > 65 years
* Informed written consent

Exclusion Criteria:

* Known amyloidosis
* Myelomatosis
* Monoclonal gammopathy of unknown significance, MGUS
* Morbus Waldenstrøm

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of cardiac amyloidosis | 1 year
  DPD scintigraphy with a Perugini Grade 2 og higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No